CLINICAL TRIAL: NCT00734084
Title: A Prospective, Non-Comparative Multi-centre Study to Evaluate the Safety and Performance of the DePuy Minimally Invasive (Preservation) Unicompartmental Knee and Instrumentation.
Brief Title: A Study to Evaluate the DePuy Minimally Invasive Unicompartmental Knee
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: After a review of status, request of investigators & since similar data was available from other sources
Sponsor: DePuy International (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT 01/34
Record Dates: First submitted 2008-08-11; First posted 2008-08-13 (Estimated); Last update posted 2015-06-09 (Estimated); Status verified 2015-06

CONDITIONS: Osteoarthritis
Keywords: Arthroplasty; Knee; UKA; Partial; Preservation
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Preservation Unicompartmental Knee (Other): Minimally invasive orthopaedic implant for single compartment knee arthritis
  Interventions: Device: Preservation Unicompartmental Knee

INTERVENTIONS:
Device: Preservation Unicompartmental Knee — Minimally invasive orthopaedic implant for single compartment knee arthritis

SUMMARY:
The primary purpose of this investigation is to evaluate the surgical performance of the DePuy Minimally Invasive (Preservation) Unicompartmental Knee and Instrumentation in a Multi-centre setting.

The secondary objective of this investigation is to evaluate the long-term survivorship of the DePuy Minimally Invasive (Preservation) Unicompartmental Knee.

DETAILED DESCRIPTION:
Primary endpoint - to demonstrate the suitability of the developed instrumentation to safely and accurately implant the preservation Unicompartmental Knee using postoperative radiographic limb and component alignment data.

Secondary endpoints - to demonstrate the survivorship and performance of the Preservation Unicompartmental Knee using the American Knee Society clinical and radiological assessment, Oxford Knee Score and survivorship analysis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, who are 40 to 75 years of age inclusive.
* Subjects who are able to give voluntary, written informed consent to participate in this investigation and from whom written consent has been obtained.
* Subjects who, in the opinion of the Investigator, are able to understand this investigation, co-operate with the investigational procedures and are willing to return to the hospital for all the required post-operative follow-ups.
* Subjects who exhibit loss of articular cartilage which is predominantly confined to a single compartment. The remaining compartments must be intact and able to bear normal loads.
* Subjects who in the opinion of the Clinical Investigator are considered to be suitable for treatment with the investigation device, according to the indications specified in the package insert leaflet.

Exclusion Criteria:

* Subjects who, in the opinion of the Investigator, have an existing condition that would compromise their participation and follow-up in this study.
* Subjects with a known history of poor compliance to medical treatment.
* Women who are pregnant.
* Subjects who are known drug or alcohol abusers or with psychological disorders that could effect follow-up care or treatment outcomes.
* Subjects who have participated in a clinical study with an investigational product in the last month.
* Subjects who are currently involved in any injury litigation claims.
* Revision of an existing unicompartmental implant.
* Subjects who have gross ligament laxity / instability.
* Subjects who have an inflammatory joint disease
* Subjects in whom there is evidence of previous joint sepsis
* Subjects who have a pre-operative flexion contracture of 15° or greater
* Subjects who have a pre-operative flexion of less than 90°
* Subjects who have a pre-operative limb deformity of greater than 15° varus or valgus
* Subjects who have morbid obesity i.e. BMI > 40%

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 247 (Actual)
Dates: Start 2001-06; Primary Completion 2004-12 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
To demonstrate the suitability of the developed instrumentation to safely and accurately implant the Preservation Unicompartmental Knee using radiographic and intra-operative assessment | 0 days
  Intraoperative

SECONDARY OUTCOMES:
To demonstrate the survivorship and performance of the Preservation Unicompartmental Knee using the American Knee Society clinical and radiographic assessment, Oxford Knee Score and survivorship analysis. | 6 months, 1, 3, 5, 10 and 15 years

CONTACTS AND LOCATIONS:
Overall Officials: Kim Dwyer, Ph.D, Study Chair — DePuy Synthes Joint Reconstruction
Locations (1):
- Sportsmed SA, 32 Payneham, Stepney, Adelaide, South Australia, Australia